CLINICAL TRIAL: NCT02056925
Title: Speckle Tracking 2D Echocardiography in Healthy Child. Comparison of Two Different Software Systems : Echopac (General Electric) and QLAB 9.0 (Philips).
Brief Title: Echocardiographic Analysis in Healthy Child.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9167
Record Dates: First submitted 2013-12-17; First posted 2014-02-06 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Healthy Child

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography

SUMMARY:
· 2D Speckle Tracking echocardiography gained importance for the evaluation of ventricle contractility. Many indications have been developed in child population. However, the comparability of measurements between different software systems is not well defined. We choose to compare two software systems very often used in paediatric subjects : Echopac by General Electric and QLAB 9.0 by Philips. We offer a randomly second echocardiography to children which have normal heart. We compare Strain and Strain rate results between the two tests with a study of variability : ultrasound variability, operator variability, reader variability.

DETAILED DESCRIPTION:
· We select children addressed to paediatric cardiologist for not serious reason (heart murmur, chest pain, sport capacity…), which had normal heart after evaluation. If they satisfied all inclusive criteria (0 to 17 years old, parental agreement, social security fund) and neither exclusive criteria (cardiac, respiratory or muscular problems, chronic diseases, drug with heart impact, poor image quality), we randomly execute a second echocardiography. Echocardiography are done with Vivid 7 ultrasound (General Electrics) and/or IE 33 ultrasound (Philips) by one or two trained operators. Strain loops are taken on three standard apical views (two, three and four-chamber views), short axis midventricular and aortic views, sub-costal short axis aortic view and sub-costal four-chamber apical views. Strain analysis are done in a second steps by one or two trained readers with adapted software : Echopac (General Electrics) or QLAB 0.0 (Philips). Strain and Strain rate results are collected for each ventricle in each dimension.We compare results between the two tests and done statistical analysis with a study of variability : ultrasound variability, operator variability, reader variability (correlation coefficient). We also done a feasibility study with use of "poor image quality"exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* child (0 to 17 years included)
* normal heart
* parental agreement
* affiliate with social security fund

Exclusion Criteria:

-

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
strain | during echocardiography
  Strain and Strain rates measurements for each ventricle in longitudinal and radial dimension with a study of variability: ultrasound variability, operator variability, reader variability

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Principal Investigator — UH Montpellier
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

REFERENCES:
- [Result] Amedro P, Bredy C, Guillaumont S, De La Villeon G, Gamon L, Lavastre K, Meli AC, Richard S, Cazorla O, Lacampagne A, Mura T, Vincenti M. Speckle tracking echocardiography in healthy children: comparison between the QLAB by Philips and the EchoPAC by General Electric. Int J Cardiovasc Imaging. 2019 May;35(5):799-809. doi: 10.1007/s10554-018-01516-2. Epub 2019 Jan 8. PMID 30623351